CLINICAL TRIAL: NCT04305652
Title: Impact of the Progressively Lowered Stress Threshold Model on Alzheimer's Patient and Caregivers' Care Outcomes: A Randomized Controlled Trial
Brief Title: The Progressively Lowered Stress Threshold Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Güler Duru Aşiret, Principal Investigator, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/248
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease; CAREGİVER
Keywords: Alzheimer Disease; Caregivers; Care satisfaction; Agitation
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Masking Description: No Intervention: Control group Experimental: Experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Care providers of Alzheimer's patients aged 65 and over (the standardized Mini-Mental State Examination (MMSE) test cognitive levels score is 19 and below )
- Experimental group (Experimental): Care providers of Alzheimer's patients aged 65 and over (the standardized Mini-Mental State Examination (MMSE) test cognitive levels score is 19 and below) The caregivers of Alzheimer's patients will be trained for 3 months according to the Progressively Lowered Stress Threshold Model with a home visit.
  Interventions: Other: The Progressively Lowered Stress Threshold Model

INTERVENTIONS:
Other: The Progressively Lowered Stress Threshold Model — PLST is a conceptual model for reducing behavioral symptoms in individuals with dementia. The PLST model provides the foundation for a psychoeducational intervention that assists formal and informal caregivers in understanding behaviors and planning care for individuals with dementia. If the model is to be applied at home, at least three home visits are made in line with the listed principles. While making a diagnosis during the first home visit, a maintenance plan for the problems is created in other home visits and the caregiver is trained to implement the care plan. After the home visits, the process is carried out by providing counseling through telephone calls or face-to-face interviews when necessary.
  Arms: Experimental group

SUMMARY:
Today, with the prolongation of human life, the elderly population has increased and the frequency of diseases seen in old age has increased due to this situation. The most common of these diseases is Alzheimer's disease. The Progressively Lowered Stress Threshold (PLST) is a conceptual model for reducing behavioral symptoms in individuals with dementia. In this study, it is aimed to determine the effect of interventions according to Decreased Stress Threshold Model on the level of neuropsychiatric symptoms and agitation of Alzheimer's patient and caregivers care satisfaction and life satisfaction.

DETAILED DESCRIPTION:
Today, with the prolongation of human life, the elderly population has increased and the frequency of diseases seen in old age has increased due to this situation. The most common of these diseases is Alzheimer's disease. Alzheimer's disease is a progressive neurodegenerative disease which causes cognitive decline and various neuropsychiatric behavioral disorders and disorders in daily living activities. The emergence of these symptoms of Alzheimer's disease leads to an increase in the costs of care provided and a great distress for caregivers. In the literature, it is recommended to use nonpharmacological approaches as the first choice in the treatment of behavioral and psychological symptoms. One of the non-pharmacological approaches is the interventions according to the Progressively Lowered Stress Threshold Model. In this method, taking into account the individuality of the patient, focusing on the interaction of the Alzheimer's patient with the environment and the rearranging of the environment for the reduction of cognitive abilities, focuses on creating a less stressful environment. Since this model uses the steps of the nursing process, home visits are made. This study will be carried out with Alzheimer's patients and caregivers from Aksaray University Education and Research Hospital's Home Health Services unit. In this study, it is aimed to determine the effect of interventions according to Decreased Stress Threshold Model on the level of neuropsychiatric symptoms and agitation of Alzheimer's patient and caregivers care satisfaction and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above,
* Caring for moderate to mild Alzheimer's patients (test cognitive levels score is 19 and below)
* Being a close relative of the patient,
* Being the primary caregiver,
* Having volunteered to participate in the study
* There is no problem with communication

Exclusion Criteria:

* Younger than 18,
* Caring for an advanced Alzheimer's patient
* Paid caregiver
* Having a communication problem

the standardized Mini-Mental State Examination (MMSE) test cognitive levels score is above 20 points

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory | 3 month
  Cohen-Mansfield Agitation Inventory, assessing the frequency of agitation symptoms.The total score that can be taken from the scale ranges between 29-203.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | 3 month
  Neuropsychiatric Inventory used to measure behavioral outcome in particular.If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
The Turkish version of the Carer's Assessment of Satisfaction Index.There was no cut-point in score interpretation, and a higher total score indicates higher caregiver satisfaction | 3 month
  CASI, assessing caregiver satisfaction.
Life Satisfaction scale | 3 month
  It evaluates the life satisfaction of caregivers.The higher the score obtained from the scale, the higher the satisfaction.
the standardized Mini-Mental State Examination | 1month
  SMMT evaluates cognitive status. Seniors with a SMMT score 19 and below (min.0 - max. 30) were included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Kütmeç Yılmaz, Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department,; Kadriye Sayın Kasar, Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department,
Locations (1):
- Aksaray University Health Science Faculty, Aksaray, Turkey (Türkiye)